CLINICAL TRIAL: NCT01682200
Title: An Open Label Pilot Clinical Trial on the Efficacy and Safety of ProOxy Facial Spray (Topical 15% Oxygen Solution) in the Treatment of Moderate Facial Acne Vulgaris Among Filipino Patients
Brief Title: Clinical Trial on the Effects and Side Effects of ProOxy in the Treatment of Acne
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medivet Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PaspaPharma-04
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Acne Vulgaris
Keywords: moderate; facial acne; acne vulgaris
MeSH Terms: conditions — Acne Vulgaris; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ProOxy, Effects and Side Effects in treating acne (Experimental): Patients are instructed to clean the face with ProOxy facial cleanser and then spray on the face wet enough but not dripping twice daily (upon waking up and before bedtime) for 3 months.
  Interventions: Drug: ProOxy

INTERVENTIONS:
Drug: ProOxy — Clean the face with ProOxy facial wash before spraying ProOxy on the face enough to wet it twice daily, upon waking up and before bedtime.
  Other Names: 15% Oxygen solution spray

SUMMARY:
This study was conducted to determine the effects and side effects of ProOxy facial spray in the treatment of acne.

DETAILED DESCRIPTION:
A study on the effects and side effects of ProOxy facial spray was done. Sixty people were selected and approved to participate in this study. Pictures of the face (frontal,left side and right side) were taken upon acceptance, during and after treatment at 4,8 and 12 weeks intervals.

ELIGIBILITY:
Inclusion Criteria:

* patients with acne on their faces only
* patients who are at least 18 years of age
* patients who have normal and disease free skin at the dorsal surface of the upper arm.
* patients who are willing to follow instructions on both the Patch Test Part one and Part Two procedures and to follow scheduled visits.

Exclusion Criteria

* patients with systemic illnesses(such as but not limited to heart disease, hypertension, diabetes, cancer, liver disease, kidney disease)
* patients with very dark skin color, Fitzpatrick skin type V-VI, who are prone to post=inflammatory hyperpigmentation.
* patients with intake of oral medications including glucocorticoids or any immuno-suppressants or who have undergone ultraviolet phototherapy for the past 2 weeks prior to the patch test.
* patients with history of contact dermatitis, dermatographism or anaphylaxis.
* patients with history of eczematous and inflammatory dermatitis, seborrheic dermatitis and psoriasis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Changes in the appearances,sizes of the acne lesions as well as the disappearance of acne on the face. | 4,8,12 weeks post application of the spray
  Upon acceptance,pictures are taken and acne lesions are identified and counted and after 4,8, and 12 weeks during and after application of ProOxy.

CONTACTS AND LOCATIONS:
Locations (2):
- Philippines (2):
  - Mary Chile General Hospital, Manila, National Capital Region
  - Far Eastern University Hospital, Dept of Family Medicine, Quezon City, National Capital Region